CLINICAL TRIAL: NCT00109577
Title: Randomized Placebo-controlled Phase II Trial of MCN36 in Adults With Bipolar Disorder
Brief Title: Clinical Trial of a Nutritional Supplement in Adults With Bipolar Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit large enough sample; large expectancy effects but no adverse events
Sponsor: University of Calgary (Other)
Collaborators: Alberta Innovation and Science (Other)
Responsible Party: Principal Investigator, Bonnie Kaplan, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18229; AIS99-03A (01406-005-23)
Record Dates: First submitted 2005-04-28; First posted 2005-04-29 (Estimated); Results first posted 2012-09-11 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; mood disorders; manic depression; nutrition
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Placebo comparator, 6 placebo capsules three times a day
  Interventions: Drug: Placebo
- 1 (Experimental): nutritional supplement intervention, 6 nutritional supplement capsules three times a day; the nutritional supplement is a 36-ingredient micronutrient supplement (primarily vitamins and minerals) and is referred to as MCN36, because it contains 36 nutrients.
  Interventions: Drug: MCN36 (nutritional supplement)

INTERVENTIONS:
Drug: MCN36 (nutritional supplement) — nutritional supplement
  Arms: 1
Drug: Placebo — nutritional supplement
  Arms: 2

SUMMARY:
The purpose of the trial was to determine whether a 36-ingredient micronutrient supplement (primarily vitamins and minerals) is beneficial for the treatment of bipolar disorder, when studied under randomized and fully blinded conditions and compared to a placebo. The supplement is referred to as MCN36, because it contains 36 nutrients. Based on the preliminary research on this supplement, it is hypothesized that patients who take MCN36 for 8 weeks will experience improved mood stability relative to those who take the placebo. All participants must live EITHER in the vicinity of Calgary, Alberta, Canada, OR in the area of San Diego, California.

DETAILED DESCRIPTION:
This RCT (randomized clinical trial) compared MCN36 to placebo in patients randomized to receive one or the other for 8 weeks. Close medical supervision was provided with weekly appointments. At the end of the 8 weeks, all participants were offered the opportunity of entering an 8-week open-label extension.

The efficacy objective of this study was to assess the efficacy of MCN36 compared with placebo in otherwise medication-free adults with bipolar disorder I and II, in improving overall symptomatology at the end of 8 weeks of therapy as assessed under randomized and fully blinded conditions

* as measured by the clinician using the Overall Bipolarity Index (OBI) (primary outcome measure).
* as measured by the clinician using the Clinical Global Impressions for Bipolar Disorder (CGI-BP) for Severity.
* as measured by self-report recorded on the Outcome Questionnaire (OQ).
* in terms of rate of response, with response defined as a reduction of 50% or more in either the depression or the mood elevation component of the OBI.
* in terms of functional states and health-related quality of life as measured by The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36).

The safety-related objective was to assess the safety of MCN36 compared with placebo in terms of

* laboratory analyses
* treatment-emergent adverse events, which will be solicited at each appointment using the Adverse Event Log.

Participants had two appointments for screening and confirming suitability for the trial. Between those two appointments, they provided a blood sample, and met with a research nurse. They also kept a 7-day food record of their food intake prior to the second appointment. If suitability was confirmed at the second visit, they entered the randomized phase.

ELIGIBILITY:
Inclusion Criteria:

* Must meet the criteria for bipolar disorder I or II as defined in DSM-IV-TR based on clinical assessment and confirmed by structured diagnostic interview (SCID-P).
* Must be symptomatic on the Hamilton Depression Scale and the Young Mania Rating Scale
* Must be free of medications or herbal/nutritional supplements with primarily central nervous system activity
* Must be able to eat at least a snack three times per day, so that the capsules will not be ingested on an empty stomach

Exclusion Criteria:

* Current or lifetime diagnosis of any of the following according to DSM-IV-TR criteria: Schizophrenia, Schizophreniform Disorder, Schizoaffective Disorder, Delusional Disorder, Psychotic Disorder Not Otherwise Specified, Delirium of any type, Dementia of any type, Amnestic Disorder, unless there is substantive reason to believe the patient was misdiagnosed.
* Alcohol dependence or abuse in the previous six months.
* Dependence or abuse of substances other than alcohol in the previous two years.
* Any Psychotic Disorder due to a General Medical Condition in the previous two years
* Hospitalization for treatment of a mental disorder within the previous 6 months.
* Current use of any other medication or herbal/nutritional supplement with primarily central nervous system activity.
* Neurological disorder involving brain or other central function.
* Severe headaches of any type (including migraine) within the previous 3 months.
* Unstable illnesses either with active significant symptoms or requiring medication changes within the previous 4 months.
* Abnormal laboratory values detected at screening, in particular an ALT or AST greater than 2 times the upper limit of normal, or creatinine greater than 1.75 times the upper limit of normal.
* Uncorrected or unstable hypothyroidism or hyperthyroidism in the previous 12 months.
* Medically diagnosed Irritable Bowel Syndrome, or any other chronic gastrointestinal problem, within the previous 3 years.
* Current or lifetime metabolic disorder or problem, such as phenylketonuria or Wilson's disease.
* A course of treatment with electroconvulsive therapy (ECT) within the previous 12 months, or a lifetime history of four or more courses of ECT.
* Current bacterial, viral, fungal, parasite or other infection.
* Women who are pregnant or breast-feeding; women of childbearing potential who are not using a medically accepted means of contraception when engaging in sexual intercourse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie J Kaplan, PhD, Principal Investigator — University of Calgary
Locations (2):
- Dr Estelle Goldstein, San Diego, California, United States
- University of Calgary Faculty of Medicine, Calgary, Alberta, Canada

REFERENCES:
- [Background] Kaplan BJ, Simpson JS, Ferre RC, Gorman CP, McMullen DM, Crawford SG. Effective mood stabilization with a chelated mineral supplement: an open-label trial in bipolar disorder. J Clin Psychiatry. 2001 Dec;62(12):936-44. doi: 10.4088/jcp.v62n1204. PMID 11780873
- [Background] Kaplan BJ, Fisher JE, Crawford SG, Field CJ, Kolb B. Improved mood and behavior during treatment with a mineral-vitamin supplement: an open-label case series of children. J Child Adolesc Psychopharmacol. 2004 Spring;14(1):115-22. doi: 10.1089/104454604773840553. PMID 15142398
- [Background] Kaplan BJ, Crawford SG, Gardner B, Farrelly G. Treatment of mood lability and explosive rage with minerals and vitamins: two case studies in children. J Child Adolesc Psychopharmacol. 2002 Fall;12(3):205-19. doi: 10.1089/104454602760386897. PMID 12427294
- [Background] Popper CW. Do vitamins or minerals (apart from lithium) have mood-stabilizing effects? J Clin Psychiatry. 2001 Dec;62(12):933-5. doi: 10.4088/jcp.v62n1203. No abstract available. PMID 11780872
- [Background] Simmons M. Nutritional approach to bipolar disorder. J Clin Psychiatry. 2003 Mar;64(3):338; author reply 338-9. doi: 10.4088/jcp.v64n0317d. No abstract available. PMID 12716280
- [Background] Kaplan BJ, Crawford SG, Field CJ, Simpson JS. Vitamins, minerals, and mood. Psychol Bull. 2007 Sep;133(5):747-60. doi: 10.1037/0033-2909.133.5.747. PMID 17723028

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Comparator: Placebo comparator capsules
- Micronutrient Formula: nutritional supplement capsules containing 36-ingredients primarily vitamins and minerals; the supplement is referred to as MCN36, because it contains 36 nutrients.
Period: Overall Study
Arm/Group | Placebo Comparator | Micronutrient Formula
Started | 20 | 20
Completed | 17 | 17
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo Comparator: Placebo comparator
- Micronutrient Formula: nutritional supplement
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator | Micronutrient Formula | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 40 (13) | 35 (9) | 37.5 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7
  Canada | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Mood as Evaluated by the Overall Bipolarity Index (Composite of the Hamilton Depression Scale and the Young Mania Rating Scale)
Description: Change in mood from baseline to final visit, as evaluated by the Overall Bipolarity Index (composite of the Hamilton Depression Scale and the Young Mania Rating Scale); minimum possible score is 0 and maximum possible score is 103; higher scores mean worse symptomatology
Time Frame: Baseline to 8 weeks
Population: All participants were included, since the analysis was intent-to-treat with last observation carried forward
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Micronutrient Formula: nutritional supplement capsules
Arm/Group | Placebo Comparator | Micronutrient Formula
Number analyzed (Participants) | 20 | 20
units on a scale | -21.1 (3.4) | -18.9 (2.9)

2. Secondary Outcome: Global Clinical Impressions
Time Frame: Baseline to 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Outcome Questionnaire --- a Self-report Questionnaire
Time Frame: Baseline to 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Medical Outcomes Study 36-Item Short Form Health Survey (SF-36)
Time Frame: Baseline to 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Placebo Comparator | Micronutrient Formula
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No